CLINICAL TRIAL: NCT03333720
Title: Compliance, Tolerance and Acceptability of a Tablet Protein Substitute for the Dietary Management of Phenylketonuria
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PKU.LP2017
Record Dates: First submitted 2017-09-18; First posted 2017-11-07 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Phenylketonurias
Keywords: Phenylketonuria; Inherited Metabolic Disorders
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Intervention is phenylalanine-free protein substitute. Following a 7 day baseline period, all recruits will receive the new phenylalanine-free protein substitute daily for 28 days in addition to routine nutritional management. The study product prescription will be specified on an individual basis by the metabolic Dietitian responsible for the patient's nutritional management and will be dependent on age, bodyweight and medical condition of the patient, but will wholly replace their currently prescribed tablet protein substitute and multivitamin supplements.
  Interventions: Dietary Supplement: Phenylalanine-free protein substitute tablets

INTERVENTIONS:
Dietary Supplement: Phenylalanine-free protein substitute tablets — Thirty eligible PKU patients (≥ 8 years), identified as current tablet users, will be recruited to this study. Patients will firstly observe a 7-day baseline period. During baseline, patients will continue with their existing diet and protein substitute prescription before receiving Phenylalanine-free protein subsitute tablets daily for 28 days in addition to appropriate nutritional management.

SUMMARY:
Thirty eligible PKU patients (≥ 8 years), identified as tablet protein substitute users, will be recruited. Patients will firstly observe a 7-day baseline period, in which participants will continue with their existing diet, protein substitute and multi vitamin prescription. Patients will then receive the phaenylalanine-free protein substitute tablets daily for 28 days in addition to appropriate nutritional management. The aim of this prospective, single arm trial is to evaluate the acceptability (compliance, tolerance and palatability) of the phenylalanine-free protein substitute tablets in patients with proven PKU. The primary outcome measure is compliance, with secondary outcome measures of gastrointestinal tolerance, acceptability, blood amino acids, dietary intake, anthropometry and safety.

DETAILED DESCRIPTION:
Protein substitutes are typically presented in powder format and reconstituted in water to a set volume, but may also be offered in ready-to-drink formats or as a gel. Notwithstanding recent advancements related to the taste, scent and texture (organoleptic properties) of commercially available protein substitutes, a small proportion of PKU patients choose to consume tablet-based protein substitutes. In this sense, anecdotal evidence suggests that in the UK approximately 80-100 PKU patients consume tablet protein substitutes. Despite the need to consume large quantities, protein substitutes in tablet format may help overcome some of the aforementioned limitations compared to powdered or ready-to-drink preparations, but also offer additional benefits including convenience and reduced preparation.

Although usage of tablet-based protein substitutes is low in comparison to powdered preparations, early evidence from MacDonald and colleagues suggests tablet protein substitutes are an equally effective strategy to manage PKU in older children, teenagers and adults. Tablet-based protein substitutes, however, only offer a balanced mixture of essential and non-essential amino acids. Considering the daily burden and discipline required to follow the restrictive low-protein diet, reports suggest achieving full compliance with tablet-based protein substitutes is difficult, and this becomes especially challenging when given alongside multi vitamin supplements. To elaborate, patients solely consuming protein substitutes in tablet format may be required to consume 70-140 tablets per day (average = 75 tablets per day) alongside an additional 5 prescribable vitamin and mineral tablets. In this instance, it may be beneficial if tablet-based protein substitutes combined amino acids with vitamins, minerals and trace elements.

At present, tablets combining amino acids with vitamins, minerals and trace elements are currently unavailable. As such, the sponsor has produced a tablet-based protein substitute designed for individuals aged 8 years and older. Developed specifically for the dietary management of proven PKU, the phenylalanine-free protein substitute tablets comprise an adapted mixture of essential and non-essential amino acids (excluding phenylalanine) and are combined with carbohydrates, DHA, vitamins and selected minerals and trace elements. As such, the aim of this intervention trial is therefore to evaluate the acceptability (compliance, gastrointestinal tolerance and palatability) of the tablets, while also capturing information related to blood amino acid profiles, dietary intake, anthropometry and safety as part of a low phenylalanine dietary regimen in PKU patients. Thirty eligible PKU patients (≥ 8 years), identified as current tablet users, will be recruited. Patients will firstly observe a 7-day baseline period. During baseline, patients will continue with their existing diet and protein substitute prescription before receiving the tablets daily for 28 days in addition to appropriate nutritional management.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 8 years of age and older
* Diagnosed with proven PKU
* Consume a minimum of 20g protein equivalent in tablet format while enrolled on to the trial
* If routine care and dietary management is not different from normal PKU care and dietary management, preconception patients may be considered
* Have written informed consent from patient or parent/carer carer

Exclusion Criteria:

* Requiring nutritional support (including enteral and parenteral nutrition)
* Major hepatic or renal dysfunction
* Maternal PKU patients (if a patient becomes pregnant during the study they will be withdrawn on immediate notice to the Metabolic Dietitian responsible for the patient's care)
* Participation in other studies within 1 month prior to entry of this study
* Investigator concern around willingness/ability of patient to comply with protocol requirements

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Daily Compliance | 35 days
  Compliance with currently prescribed protein substitute and prescribed multivitamin supplements will be assessed daily from days 1-7 and recorded as a percentage of tablets consumed comapred to prescription (0-100%). Compliance with the study product will subsequently be assessed daily from days 8-35. Compliance throughout the trial will be assessed using standarised questionnaires, where patients document number of med versus number of tablets prescribed. A percentage compliance level based on per patient and total patients will be computed to define overall compliance where a higher percentage represents better overall compliance.

SECONDARY OUTCOMES:
Treatment-Emergent tolerability | 12 days
  Gastrointestinal tolerance (including diarrhoea, constipation, nausea, vomiting, abdominal pain, bloating, flatulence and burping) will be assessed via questionnaire using the scale (absent, mild, moderate, severe).
Patient Acceptability | 2 days
  Acceptability (ease of use and palatability) will be assessed via questionnaire.
Metabolic control | 2 days
  Blood phenylalanine, blood tyrosine and other amino acids. Fingertip-capillary blood samples will be collected in the fasted state at baseline observations (day 1), and on the last day of the intervention period (day 35). Collected samples will be analysed for blood phenylalanine, tyrosine and 16 other proteinogenic amino acids, 2 non-proteinogenic amino acids and 1 amino sulfonic acid.
Nutritional Intake | 2 days
  To assess habitual dietary intake, 24 hour dietary recalls will be completed during baseline and at the end of the intervention period.
Weight | 2 days
  Measures of weight (kg) will be made during baseline observations and at the end of the intervention period.
Height | 2 days
  Measures of weight (kg) will be made during baseline observations and at the end of the intervention period.
Incidence of study product emergent adverse events [safety]. | Baseline
  All adverse events will be recorded throughout the study (as and when they occur). Consequently, there is no specific time frame as the frequency of adverse events can not be predicted.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stratton, PhD, Study Director — Nutricia, Inc.

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.